CLINICAL TRIAL: NCT01124578
Title: Validate the Acceptability of Egret's Extended Use Product as Compared to the Existing Daily Change-out Product
Brief Title: Study the Average Aerobic Bioburden Levels on Catheters After Use With Egret Catheter and the Predicate Device
Status: Completed | Type: Observational
Sponsor: Egret Medical Products Inc. (Industry)
Responsible Party: David Barton, BA, RRT, RCP, Medical City Dallas Hospital
Other Study IDs: RT 2008-001
Record Dates: First submitted 2010-05-07; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Suction Catheter Bioburder Level After Patient Use.
Keywords: Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Existing used daily change-out device
- Egret: Extended Use Catheter w/BIOSAFE

SUMMARY:
PURPOSE OF EVALUATION: This study will verify & validate the acceptability of Egret's extended use product as compared to the existing daily change-out product. Based on an extensive in-vitro study, Egret's product confirmed significant kill for both positive and negative gram bacteria. In addition to meeting all of the current product requirements, total aerobic bio-burden on the catheters will be tested at various intervals for up to 10 days of use. The current used product will be used as a control group that is to be changed out daily as per current policy. The control group will be tested for total aerobic bacteria counts on the last day of use.

DETAILED DESCRIPTION:
Protocol

Title: Extended Use In-line Endotracheal Suction Catheter w/BIOSAFE

Protocol Number: RT 2008-001

Study Director: Richard C. Dowdy

Study Director's Address and Method of Contact:

Egret Medical Products Inc. Richard C. Dowdy 2713 Industrial Lane Garland, TX 75041 (214) 291-0238 Phone (817) 991-7459 Cell (214) 291-0243 Fax rdowdy@egretmedical.com

I. PURPOSE OF EVALUATION: This test will verify & validate the acceptability of Egret's extended use product as compared to the existing Ballard's daily change-out product. In addition to meeting all of the current product requirements, total aerobic bio-burden on the catheters will be tested at various intervals for up to 10 days of use.

II. BACKGROUND: Prior to this evaluation, a baseline study was conducted at Medical City to determine the existing total aerobic bio-burden after one day of use, using 25 randomly selected Ballard catheters as per the attached protocol. The data from the baseline study were used to establish an appropriate sample size for the Extended Use Protocol. This data gathered under this Extended Use Protocol will be compared to the baseline data to determine the effectiveness of Egret's antimicrobial properties during extended use.

III. POTENTIAL RISK TO PATIENT: Closed endotracheal suction catheters are intended to maintain a hermetical seal. However, such catheters have a propensity to build up bio- film on the tip area and require saline rinsing and cleaning after use. Egret's catheter is compounded with a non-leaching antimicrobial to address this issue. There is the possibility that excessive patient secretions can over saturate any closed suction catheter. Egret has addressed this concern by incorporating a unique squeegee-and-filter design that facilitates tip cleaning and prevents debris from migrating from the cleaning chamber to the sleeve area.

IV. BENEFTS OF THE EGRET MEDICAL DEVICE

1. The catheter contains a non-leaching antimicrobial agent that enables product to be used safely for up to fourteen (10) days.
2. Based on previous in-vitro testing, the Egret product with BIOSAFE has been found to reduce bacteria counts over extended time.
3. Minimizing the frequency of change-out of the closed catheter system will reduce the chance for cross-contamination since the air way will be opened less frequently, e.g., every five days versus daily.
4. Less frequent product change-out reduces the need to manipulate the ET-Tube. The more the ET-Tube is manipulated, the greater the chance upper airway contents trapped above the cuff can enter the pulmonary bed.
5. The catheter reduces bacteria colonization over the span of its use
6. The swivel connector enables accessories to be easily connected and disconnected.
7. An integrated positive lock valve facilitates use and prevents gas from escaping when not in use.
8. A uniquely designed filter is incorporated into the device's manifold that provides a 95% BFE level to prevent cross-contamination to caregiver and patient.
9. Egret's devices are MRI safe - no metal parts are used in assembly.

V. PRODUCT to BE EVALUATED:

Product Code Description Size 454 Egret 14 Fr. T-Piece - Extended use 14 FR/4.6 mm 54 cm (21.75") length

VI. INVESTIGATOR David Barton, BA, RRT, RCP

VII. SPONSOR Egret Medical Products Inc.

VIII. AFFLICATION OF APPLICANT Egret Medical Products Inc.

IX. FUNDING AGIENCIES Egret Medical Products Inc.

X. ANTICIPATED TEST DATES April 2008-May 2008

XI. METHODOLOGY:

1. Egret will provide 100 units of product to support use testing requirements
2. An in-service meeting will be held by Egret facilitators prior to beginning the test to ensure participants are aware of the use test requirements and responsibilities.
3. During the test period, the Egret product will be used instead of the specific normally used for the procedure for up to 10 days if needed.
4. This device is to be used per existing Medical City Policy RCSCC12 with the exception that change- out is not required daily, and that the Egret device can be used up to 10 days or until extubation.
5. Careful instruction is to be given the caregiver on how catheter is to be flushed and rinsed after suctioning. This step is essential to maintain the patency of the catheter as well as to reduce bio- burden that the catheter must combat.
6. Clinical Trial Subject Tracking - As per the attached spreadsheet, product installation and usage is to be tracked by the investigator. Products provided from Egret will be discreetly numbered 1 thru 100 on the bottom of each suction catheter valve.
7. Arrangements have been made with MicroChem Laboratory, Inc. to conduct total aerobic bio-burden using the same the method used for the baseline study.
8. After product has been used, representative samples are to be red bagged and sent by courier to MicroChem to conduct aerobic bacterial testing. Transportation and testing requirements are clearly outlined in an approved test protocol.
9. Egret personnel will be present at Medical City to facilitate and observe the use of the test product for the duration of the test period.
10. At the completion of the test period, healthcare participants will complete a questionnaire concerning the Egret use test product as compared to the existing Ballard product.
11. All test products at the end of the test period will be return to Egret.
12. During the evaluation, if a caregiver perceives defect or failure, the caregiver is to contact the investigator for assessment. Products that are perceived as defective are to be set aside for additional evaluation by Egret.

XII. DATA TO BE COLLECTED: After product has been used, the healthcare participants will complete a written questionnaire concerning the test device as per attached.

XIII. DELIVERY OF PRODUCT: Available test product will be delivered to use-test site as per Medical City instructions.

XIV. RECOVERY OF PRODUCT: The investigator will be responsible for gathering all unused test product and returning it to Egret.

XV. SPECIAL INSTRUCTIONS: Participants will be briefed on the specific features of Egret's extended use product to be tested at their facility.

XVI. TEST FACILITATORS: Egret will provide on-site qualified personnel to assist with resources as required by Medical City.

XVII. APPROVALS

Study Director: Richard C. Dowdy Date: Title: Vice President

The Study Director is responsible for ensuring that no data for use in the Final Report (Outputs) has been generated before protocol approval.

Approvers: Egret Medical Products Inc. Management

Signature(s) indicate that this protocol has been reviewed and understood in its entirety and meets all criteria specified in Section 4.1, Protocol Design and Approval Policy.

Approver: Date: Title:

Approver: Date: Title:

Approver: Date: Title:

Upon approval of the protocol, the original is to be filed at the administrative offices of Egret Medical Products Inc. The study director should retain a copy of the protocol until the report is completed

Endotracheal Suctioning Catheter Use Test Questionnaire

Clinician's Name: Date:

Where Used: Oral Intubation 0 or Trach 0

Product usage questions Not Same as Improved Acceptable Current Use of Change-out label

0 0 0

Connection to suction tubing

0 0 0

Suction Valve - Ease of use

0 0 0

Gauge and feel of sheath material

0 0 0

Valve Locking Safety Feature

0 0 0

Ease of connection to trach or ET tube

0 0 0

Catheter positioning and ease of manipulation

0 0 0

Communication\visibility of depth markings

0 0 0

Use of saline port

0 0 0

Tip cleaning process and result

0 0 0

Product flexibility to prevent unnecessary ET movement?

0 0 0

Did sheath remain clean and dry? 0 0 0

Affect of heat on product function? 0 0 0

Perceived weight of product 0 0 0

Comfort to patient

0 0 0

Did end cap remain secure?

0 0 0

Ease of disconnect after use?

0 0 0

Did this product meet your expectation? 0 0 0

Additional Comments:

Thank you for your help

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to consent.

Exclusion Criteria:

* Patients who do not agree to consent or with confirmed Ventilator-associated Pneumonia (VAP)are to be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Medical City who require ventilation
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Measure total aerobic bioburden levels after patient use | 1 to 10 days
  Compare the average aerobic bio-burden level on the extended use Egret catheter to the existing used one day product after clinical use. The Egret catheter was used continuously for up to 10 days.

SECONDARY OUTCOMES:
No unexpected adverse events | 1-10 days
  Verify that there were no unexpected adverse events associated with the Egret extended use catheter.
Design Ease of Use | 1-10 days
  Obtain feedback from the respiratory care practitioners regarding comparative ease-of-use and design feature preferences between the Egret catheter and the Ballard catheter.

CONTACTS AND LOCATIONS:
Overall Officials: David Barton, BA, RRT, RCP, Principal Investigator — Medical City Hospital, Dallas, TX
Locations (1):
- Medical City Dallas Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] 1.Medical City Dallas Hospital, Policies and Procedures, Policy No. RSCC12 - Endotracheal Suctioning 2.MicroChem Labs - A Study to Measure the Total Aerobic Bacteria on Ballard Suction Catheters During 24 Hours Use with Respiratory Care Patients. This study was conducted to establish a baseline bio-burden count of catheter tips after use. 3.Nelson Laboratories - Bacterial Filtration Efficacy, Report No. 413451. This test was preformed to determine the bacterial filtration efficacy of the filter as per ASTM F2101. 4.Micro-Chem Labs - Evaluation of the Antimicrobial Properties of Sterilized and Non-Sterilized Egret Catheters Versus a Non-Treated Control Catheter During Extended Exposure to S. aureus, P. aeruginosa, and K. pneumoniae.